CLINICAL TRIAL: NCT04135053
Title: A Human Controlled Infection Study to Assess Safety, Colonisation and Immunogenicity Following Nasal Inoculation With Reconstituted Lyophilised Wild Type Neisseria Lactamica
Brief Title: A Controlled Study to Assess Safety, Colonisation and Immunogenicity of Reconstituted Lyophilised Neisseria Lactamica
Acronym: Lac5-Nasal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Lac5-Nasal
Record Dates: First submitted 2019-09-27; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Meningitis, Bacterial
Keywords: meningitis; healthy volunteer
MeSH Terms: conditions — Meningitis, Bacterial; Meningitis

STUDY DESIGN:
Intervention Model Description: A prospective dose ranging human challenge study. Nasal inoculation with reconstituted, previously lyophilised Neisseria lactamica with dose escalation / de-escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Challenge (Experimental): Challenge participants will inoculated intranasallly with reconstituted lyophilised Neisseria lactamica (lyoNlac). The initial dose will be 10^5 colony-forming units (CFU) and will be escalated or de-escalated by 1/2 - 1 log depending upon the proportion of volunteers colonies with viable N. lactamica.
  Interventions: Biological: Lyophilised Neisseria lactamica

INTERVENTIONS:
Biological: Lyophilised Neisseria lactamica — Previously lyophilised Neisseria lactamica will be reconstituted and intranasally given to participants

SUMMARY:
This study is part of a series of projects to develop and test new vaccines for meningitis. Previously researchers have given nose drops containing N. lactamica to over 350 volunteers, and shown that many of them (35-60%) can become colonised with N. lactamica and become resistant to becoming colonised with N.meningitidis without causing any illness or disease. In the future the study team would like to find out how N.lactamica helps children resist N.meningitidis, and develop new vaccines that exploit that mechanism.

DETAILED DESCRIPTION:
In this pilot research, the research team will develop and validate a modification of the methodology previously used in another UK-based human challenge experiments. The research to be conducted in this study will inform the study team whether intranasal inoculation of reconstituted lyophilised Nlac (hereafter, lyoNlac), can result in immunising colonisation of participants and the optimal dose to achieve this.

Previous challenges have been conducted using frozen stocks of Nlac but this is relatively unsatisfactory because of instability of frozen stocks, and will not be practical in Mali. The facility to reconstitute dry powdered lyoNlac into water and inoculate as a nose drop will greatly simplify the experimental method. However, it is not known whether lyoNlac can be inoculated directly into volunteers and induce successful colonisation.

In summary this is a pilot study of the safety, efficacy and immunogenicity of the intranasal inoculation of healthy human volunteers with lyoNlac. This study will determine the efficacy of lyoNlac as an agent for inducing nasopharyngeal colonisation with this organism, which is an important methodological development for ease of administration of Nlac in experimental human challenge studies. The study team will aim to determine the dose of inoculum required to induce colonisation in 80% of volunteers (the Standard Inoculum or SI). This SI will be used in future studies aiming to optimise duration of colonisation and immunogenicity induced by lyoNlac.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years inclusive on the day of enrolment
* Fully conversant in the English language
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Provide written informed consent to participate in the trial
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and inoculation
* TOPS registration completed and no conflict found

Exclusion Criteria:

* Current active smokers defined as having smoked a cigarette or cigar in the last four weeks
* N. lactamica or N. meningitidis detected on throat swab or nasal wash taken at screening
* Individuals who have a current infection at the time of inoculation
* Individuals who have been involved in other clinical trials involving receipt of an investigational product over the last 12 weeks or if there is planned use of an investigational product during the study period
* Individuals who have previously been involved in clinical trials investigating meningococcal vaccines or experimental challenge with N. lactamica
* Use of systemic antibiotics within the period 30 days prior to the challenge
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the inoculum, specifically soya.
* Contraindications to the use of ciprofloxacin, specifically a history of epilepsy, prolonged QT interval, hypersensitivity to quinolones or a history of tendon disorders related to quinolone use
* Any clinically significant abnormal finding on clinical examination or screening investigations
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data, for example recent surgery to the nasopharynx
* Occupational, household or intimate contact with immunosuppressed persons
* Pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Via the hospital Pathology service, analyse the haematology blood results of healthy volunteers inoculated with reconstituted lyophilised wild type Neisseria lactamica, taken at specified time points. | 1 year
  Blood samples will be taken at standardised visits. Results will be compared to those results collected from baseline and pre-inoculation visits. Any change in results will be recorded and, if deemed required by the medical team, further tests requested. Standard tests haematology- haemoglobin - g/L,
Via the hospital Pathology service, analyse the White Cell Count of healthy volunteers inoculated with reconstituted lyophilised wild type Neisseria lactamica, taken at specified time points. | 1 Year
  Blood samples will be taken at standardised visits. Results will be compared to those results collected from baseline and pre-inoculation visits. Any change in results will be recorded and, if deemed required by the medical team, further tests requested. Standard tests include haematology - White Cell Count - x10^9/L
Via the hospital Pathology service, analyse the Platelet Count of healthy volunteers inoculated with reconstituted lyophilised wild type Neisseria lactamica, taken at specified time points. | 1 Year
  Blood samples will be taken at standardised visits. Results will be compared to those results collected from baseline and pre-inoculation visits. Any change in results will be recorded and, if deemed required by the medical team, further tests requested. Standard tests include haematology - Platelet Count - x10^9/L
Via the hospital Pathology service, analyse the Biochemistry results of healthy volunteers inoculated with reconstituted lyophilised wild type Neisseria lactamica, taken at specified time points. | 1 Year
  Blood samples will be taken at standardised visits. Results will be compared to those results collected from baseline and pre-inoculation visits. Any change in results will be recorded and, if deemed required by the medical team, further tests requested. Standard tests include Biochemistry - Sodium - mmol/L
Via the hospital Pathology service, analyse the CRP results of healthy volunteers inoculated with reconstituted lyophilised wild type Neisseria lactamica, taken at specified time points. | 1 Year
  Blood samples will be taken at standardised visits. Results will be compared to those results collected from baseline and pre-inoculation visits. Any change in results will be recorded and, if deemed required by the medical team, further tests requested. Standard tests include Biochemistry - C-reactive protein - mg/L

SECONDARY OUTCOMES:
The dose of lyophilised Neisseria lactamica required for nasopharyngeal colonisation in 80% of inoculees. | 1 year
  The dose will be confirmed by nasal swabs and nasal washes taken from participants and analysed for bacteria by CFU counts. The desired dose will be confirmed when 80% of participants are colonised.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Read, Principal Investigator — University of Southampton
Locations (1):
- NIHR Southampton Clinical Research Facility, Southampton, United Kingdom

REFERENCES:
- [Derived] Gbesemete DF, Haidara F, Laver JR, Ibrahim M, MacLennan J, Dale AP, Gorringe AR, Traore Y, Diallo F, Badji H, Traore A, Onwuchekwa U, Jones E, Webb C, Guy J, Theodosiou AA, Faust SN, Sow SO, Heyderman RS, Tapia MD, Read RC. Controlled Human Infection of Healthy Adults With Lyophilized Neisseria lactamica Induces Asymptomatic, Immunogenic Nasopharyngeal Carriage in the United Kingdom and Mali. Open Forum Infect Dis. 2026 Jan 7;13(1):ofaf809. doi: 10.1093/ofid/ofaf809. eCollection 2026 Jan. PMID 41574175